CLINICAL TRIAL: NCT02253875
Title: A Single-centre, Open-label Study in Healthy Adult Volunteers to Determine the Effects of Multiple-dose Omeprazole (ANTRA® 40 mg qd) on the Single-dose Pharmacokinetics of Tipranavir 500 mg Coadministered With Ritonavir 200 mg
Brief Title: Study to Determine the Effects of Multiple-dose Omeprazole on the Single-dose Pharmacokinetics of Tipranavir (TPV) Coadministered With Ritonavir (RTV) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.84
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Omeprazole

ARMS (1):
- TPV + RTV + Omeprazole (Experimental)
  Interventions: Drug: Tipranavir (TPV); Drug: Ritonavir; Drug: Omeprazole

INTERVENTIONS:
Drug: Tipranavir (TPV)
  Other Names: (Aptivus ®)
Drug: Ritonavir
  Other Names: (Norvir-SEC®)
Drug: Omeprazole
  Other Names: (Antra®)

SUMMARY:
Study to determine the effects of multiple-dose omeprazole on the single-dose pharmacokinetics of tipranavir and ritonavir

ELIGIBILITY:
Inclusion Criteria:

1. Male and female healthy volunteers between 18 and 60 years of age inclusive
2. Clinically normal medical history
3. Clinically normal findings on physical examination
4. Clinically normal laboratory values
5. Body Mass Index (BMI) between 18.5 and 30 kg/m2 inclusive
6. Ability to swallow large capsules without difficulty
7. Capable of comprehending and communicating effectively with the investigator and site staff
8. Signed and dated written informed consent form, in accordance with Ethics Committee and regulatory guidelines prior to trial participation
9. Willingness to abstain from ingesting substances which may alter plasma drug levels by interactions with the cytochrome P450 system during the 14 days of the study
10. Willingness to abstain from alcohol for 48 hours prior to Visit 2 and for the duration of the study
11. Willingness to abstain from ingesting grapefruit and grapefruit juice for 7 days before Visit 2 and for the duration of the study
12. Negative pregnancy test (β-hCG)
13. Negative HIV serology
14. Negative hepatitis serology

Exclusion Criteria:

1. Any clinically significant disease (a significant disease is defined as a disease, which in the opinion of the investigator may either put the subject at risk because of participation in the study, or a disease which may influence the results of the study or the subject's ability to participate in the study)
2. Clinically significant abnormal baseline hematology, blood chemistry or urinalysis findings normal at Visit 2
3. Serum Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), cholesterol, triglyceride or glucose greater than the upper limit of normal at Visit 2
4. Treatment with any investigational drug within 90 days prior to the first dose of study medication
5. Inability to adhere to the requirements of the protocol as assessed by the investigator
6. Prior TPV use
7. Subjects who are taking or have taken medications metabolized through the Cytochrome P-450 (CYP450) enzyme system within 30 days prior to Visit 2
8. Subject with a seated systolic blood pressure either <100 mmHg or >150 mmHg; resting heart rate either <50 beats/min or >100 beats/min
9. Subject with a history of any illness or allergy that in the investigator opinion might confound the results of the study, or pose additional risk to the subject with the administering of TPV/r or omeprazole
10. Subject who have had an acute illness within 14 days prior to Visit 2
11. Subject who are currently taking or have taken over-the-counter medications in the 14 days prior to Visit 2, or subjects who are currently taking any prescription medication
12. Known hypersensitivity to TPV, RTV, omeprazole or antiretroviral drugs (marketed or experimental use as part of clinical research studies)
13. Female subjects who are of reproductive potential and who are:

    * Pregnant or breast-feeding
    * Have a positive serum β-hCG (pregnancy test) at screening visit (Visit 1)
    * Have not been using a barrier contraceptive method for at least 60 days prior to Study Day 1
    * Are not willing to use a reliable method of double-barrier contraception during the trial and for 30 days after completion or termination of the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-11; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum plasma concentration of Tipranavir in plasma) | up to 72 hours after drug administration
AUC0-72h (Area Under Plasma Concentration-time curve of Tipranavir from 0-72 hr) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
Cmax (Maximum plasma concentration of Ritonavir in plasma) | up to 72 hours after drug administration
AUC0-72h (Area Under Plasma Concentration-time curve of Ritonavir from 0-72 hr) | up to 72 hours after drug administration
AUC0-∞ (Area Under Plasma Concentration-time curve from 0 to infinity) | up to 72 hours after drug administration
MRT (Mean residence time) | up to 72 hours after drug administration
t1/2 (apparent terminal halflife) | up to 72 hours after drug administration
Tmax (Time to maximum concentration of the analyte in plasma) | up to 72 hours after drug administration
CL/F (Oral clearance) | up to 72 hours after drug administration
Vz/F (Apparent volume of distribution during the terminal elimination phase divided by the bioavailability factor) | up to 72 hours after drug administration
Number of subjects with adverse events | up to 24 days